CLINICAL TRIAL: NCT05951673
Title: Adolescent Girls Initiative for Learning and Empowerment: Impact Evaluation of a Safe Space-Based Life Skills Training and Digital Literacy Training in Nigeria
Brief Title: Adolescent Girls Initiative for Learning and Empowerment: Impact Evaluation of a Safe Space-Based Life Skills Training and Digital Literacy Training in Nigeria Space-Based Life Skills Training and Digital Literacy Training in Nigeria
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: World Bank (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AGILE IE
Record Dates: First submitted 2023-07-10; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Adolescent Behavior; Life Skills; Digital Skills; Sexual and Reproductive Health; Earning Outcomes
MeSH Terms: conditions — Adolescent Behavior; Coitus

STUDY DESIGN:
Intervention Model Description: Enrolled participants are randomized to Treatment 1 (Life skills only) Treatment 2 (Life skills + digital skills) and control group (No intervention).
Who Masked: Outcomes Assessor
Masking Description: Randomized using computer-generated randomization; Outcome assessors blinded against treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment 1 - Receives Safe Space based life skills training program (Experimental): Adolescent girls in this group receive a safe space-based life skills training program within their school.
  Interventions: Other: Safe Space based life skills training program
- Treatment 2 - Recieves Safe Space based life skills training program + digital literacy training (Experimental): Adolescent girls in this group receive a safe space-based life skills training program and a digital literacy training program within their school.
  Interventions: Other: Safe Space based life skills training program; Other: Safe Space based life skills training program + Digital Skills
- Control - No intervention (No Intervention): Adolescent girls in this group receive neither the safe space-based life skills training program nor the digital literacy training program.

INTERVENTIONS:
Other: Safe Space based life skills training program — This is a Safe Space based life skills training program given to adolescent girls. Girls receive a 12 month long training on life skills such as negotiation skills, communication skills, sexual and reproductive health, gender-based violence and climate change.
  Arms: Treatment 1 - Receives Safe Space based life skills training program; Treatment 2 - Recieves Safe Space based life skills training program + digital literacy training
Other: Safe Space based life skills training program + Digital Skills — This is a Safe Space based life skills training program given to adolescent girls complemented with a digital literacy training program. Girls receive a 12 month long training on life skills such as negotiation skills, communication skills, sexual and reproductive health, gender-based violence and climate change. The adolescent girls in this group also receive a digital literacy training program that covers content on word processing. database management and analysis, online marketing, online safety and programming.
  Arms: Treatment 2 - Recieves Safe Space based life skills training program + digital literacy training

SUMMARY:
The investigators will conduct a cluster randomized controlled trial in secondary schools in Nigeria to evaluate the impact of school-based life skills training delivered in safe spaces with and without digital literacy training. This study aims to estimate the causal impacts of the training on adolescents' school performances and retention, socio-emotional skills, digital skills, health, marriage, fertility, and labor market outcomes.

DETAILED DESCRIPTION:
This study will evaluate the impact of a safe-space based life skills training program as well as a combination of life skills and digital literacy training programs on adolescent girls' empowerment, education, economic and sexual and reproductive health outcomes. The interventions form two sub-components of the Adolescent Girls' Initiative for Learning and Empowerment project. The interventions will be delivered to secondary school girls in Northern Nigeria.

The study will be conducted in the Kaduna, Katsina and Kano states of Nigeria. The study has a randomized controlled trial research design where schools are randomly allocated to three groups. Girls in schools assigned to the first treatment group will receive the safe-space based life skills training program. Schools allocated to the second treatment group will deliver a digital literacy training program along with a safe-space based life skills training program. The third group of schools will receive neither training program until the completion of the study. Girls between the age of 15 - 20 form the target group of the study.

The study will evaluate the impact of (i) a safe space-based life skills training program on adolescent girls' empowerment, education, economic and sexual and reproductive health outcomes; and (ii) a combination of a safe-space based life skills and digital literacy training programs on adolescent girls' empowerment, education, economic and sexual and reproductive health outcomes.

A total of 8,463 girls are drawn from 273 schools in the three states. The study will conduct baseline, midline and endline surveys by interviewing the girls and their respective caregivers. The baseline survey is conducted before the intervention roll-out. The midline survey will be conducted six months after intervention completion, while the endline survey will be conducted two years after the completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in study schools
* Enrolled in Senior Secondary 1 level
* Parental consent

Exclusion Criteria:

-

Ages: 15 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8463 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
High school graduation | 24 months post intervention
  a binary indicator coded to 1 if a girl has obtained a high school diploma
School retention | 6 months post intervention
  a binary indicator coded to 1 if a girl is in school based on school registers
Marriage | 6 months post intervention
  a binary indicator coded 1 if an adolescent girl has ever been married (including cohabitation) and 0 otherwise.
Marriage | 24 months post intervention
  a binary indicator coded 1 if an adolescent girl has ever been married (including cohabitation) and 0 otherwise.
Engagement in non-farm income generating activities | 6 months post intervention
  a binary indicator coded 1 if a girl engaged in any paid non-farm activity in the last completed month
Engagement in non-farm income generating activities | 24 months post intervention
  a binary indicator coded 1 if a girl engaged in any paid non-farm activity in the last completed month
Digital financial literacy | 6 months post intervention
  a composite score based on 30 items that measure respondent's financial literacy and access to digital tools, with a higher score indicating greater literacy and access
Digital financial literacy | 24 months post intervention
  a composite score based on 30 items that measure respondent's financial literacy and access to digital tools, with a higher score indicating greater literacy and access
Socio-emotional skills index | 6 months post intervention
  a composite score based on indices that measure different socio-emotional skills, e.g., personal initiative, negotiation, decision-making, and communication
Socio-emotional skills index | 24 months post intervention
  a composite score based on indices that measure different socio-emotional skills, e.g., personal initiative, negotiation, decision-making, and communication

SECONDARY OUTCOMES:
Goal setting capacity | 6 months post intervention
  a composite score based on 8 items that measure the respondent's ability to set a goal
Goal setting capacity | 24 months post intervention
  a composite score based on 8 items that measure the respondent's ability to set a goal
Aspiration - education attainment | 6 months post intervention
  a variable that indicates the level of formal education the respondent would like to complete
Aspiration - education attainment | 24 months post intervention
  a variable that indicates the level of formal education the respondent would like to complete
Knowledge of climate change | 6 months post intervention
  a composite score calculated based on the correct answers to a list of questions related to climate change
Knowledge of climate change | 24 months post intervention
  a composite score calculated based on the correct answers to a list of questions related to climate change
Digital skills and knowledge | 6 months post intervention
  a composite score based on 31 items that measure respondent's technical and operational skills, information navigation and processing skills, communication and interaction skills, and content creation and production skills
Digital skills and knowledge | 24 months post intervention
  a composite score based on 31 items that measure respondent's technical and operational skills, information navigation and processing skills, communication and interaction skills, and content creation and production skills
Knowledge of productivity program | 6 months post intervention
  a composite score of items developed based on the digital literacy training curriculum
Knowledge of productivity program | 24 months post intervention
  a composite score of items developed based on the digital literacy training curriculum
School engagement | 6 months post intervention
  a composite score based on 8 items that measure respondent's school engagement
School absenteeism | 6 months post intervention
  number of days a girl missed in the last completed month
Enrollment in tertiary education | 24 months post intervention
  a binary indicator coded to 1 if a girl is enrolled in tertiary education
Sexual violence | 6 months post intervention
  a composite score based on the frequency of different types of sexual violence reported by the respondent
Sexual violence | 24 months post intervention
  a composite score based on the frequency of different types of sexual violence reported by the respondent
Bullying | 6 months post intervention
  a composite score based on the frequency of different types of bullying reported by the respondent
Bullying | 24 months post intervention
  a composite score based on the frequency of different types of bullying reported by the respondent
Knowledge on school-related gender-based violence | 6 months post intervention
  the fraction of correct responses to 12 questions that ask whether an act is considered violence
Knowledge on school-related gender-based violence | 24 months post intervention
  the fraction of correct responses to 12 questions that ask whether an act is considered violence
Gender attitudes and beliefs | 6 months post intervention
  a composite score for (a) gender equality beliefs based on the frequency of the different types of favorable gender equality beliefs, and (b) acceptability of IPV based on the frequency of the different types of violence girls find acceptable
Gender attitudes and beliefs | 24 months post intervention
  a composite score for (a) gender equality beliefs based on the frequency of the different types of favorable gender equality beliefs, and (b) acceptability of IPV based on the frequency of the different types of violence girls find acceptable
Pregnancy | 6 months post intervention
  a binary indicator coded 1 if an adolescent girl has ever been pregnant and 0 otherwise.
Pregnancy | 24 months post intervention
  a binary indicator coded 1 if an adolescent girl has ever been pregnant and 0 otherwise.
Sexual behavior - ever had sex | 6 months post intervention
  a binary indicator coded 1 if an adolescent girl has ever had sex and 0 otherwise.
Sexual behavior - ever had sex | 24 months post intervention
  a binary indicator coded 1 if an adolescent girl has ever had sex and 0 otherwise.
Drug use - ever used drug | 6 months post intervention
  a binary indicator coded 1 if an adolescent girl has ever used drugs and 0 otherwise
Drug use - ever used drug | 24 months post intervention
  a binary indicator coded 1 if an adolescent girl has ever used drugs and 0 otherwise
Health knowledge | 6 months post intervention
  a composite score for (a) correct answers on knowledge of SRH, menstruation, and puberty, and (b) correct answers on knowledge of nutrition
Health knowledge | 24 months post intervention
  a composite score for (a) correct answers on knowledge of SRH, menstruation, and puberty, and (b) correct answers on knowledge of nutrition
Sector - ICT | 24 months post intervention
  a binary indicator coded 1 if a girl engages in income-generating activities related to ICT
Number of days worked | 6 months post intervention
  number of days a girl was engaged in paid work in the last complete month
Number of days worked | 24 months post intervention
  number of days a girl was engaged in paid work in the last complete month
Income | 6 months post intervention
  aggregate income earned in the last completed month
Income | 24 months post intervention
  aggregate income earned in the last completed month
Savings | 6 months post intervention
  amount saved in the last completed month
Savings | 24 months post intervention
  amount saved in the last completed month
Perceived social support | 6 months post intervention
  mean score from the Multidimensional Scale of Perceived Social Support
Perceived social support | 24 months post intervention
  mean score from the Multidimensional Scale of Perceived Social Support

CONTACTS AND LOCATIONS:
Overall Officials: Lea Rouanet, PhD, Principal Investigator — World Bank
Locations (1):
- World Bank Group, Abuja, Nigeria

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data outside the team to ensure participants' privacy.